CLINICAL TRIAL: NCT06681493
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and PK/PD of YZJ-4729 Tartrate Injection After A Single Ascending Dose
Brief Title: A Phase 1 Study of YZJ-4729 Tartrate Injection in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YZJ-4729-1-01
Record Dates: First submitted 2024-10-31; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Analgesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Part A Experimental: YZJ-4729 Tartrate injection; Part A Control: YZJ-4729 simulated injection
  Interventions: Drug: YZJ-4729 Tartrate injection; Drug: YZJ-4729 simulated injection
- Part B (Experimental): Subjects will receive YZJ-4729 Tartrate injection
  Interventions: Drug: YZJ-4729 Tartrate injection

INTERVENTIONS:
Drug: YZJ-4729 Tartrate injection — Infusion, QD
Drug: YZJ-4729 simulated injection — Infusion, QD
  Arms: Part A

SUMMARY:
Part A

Primary objective:

• To evaluate the safety, tolerability, and pharmacokinetic profile of a single dose of YZJ-4729 tartrate injection.

Secondary objectives:

* To investigate the PK/PD profile of YZJ-4729 tartrate injection administered as a single dose;
* To investigate the metabolic transformation characteristics of YZJ-4729 tartrate;
* To assess the relationship between plasma concentrations and change in QT interval (C-QT) and the effect on QT interval in subjects after a single dose of YZJ-4729 tartrate injection.

Part B

Primary objective:

• To evaluate the safety, tolerability and pharmacokinetic profile of YZJ-4729 tartrate injection administered at the same dose and at different infusion rates .

Secondary objectives:

• To investigate the PK/PD profile of YZJ-4729 tartrate injection administered at the same dose and at different infusion rates.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged between 18 and 45 years (inclusive) on the day of signing the informed consent;
2. Male subjects weighing no less than 50 kg and female subjects weighing no less than 45 kg. Body mass index within the range 19.0-26.0 kg/m 2 (inclusive);
3. Subjects in good health without a history of serious diseases and chronic diseases such as respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system and mental system;
4. From the date of signing the informed consent form until 6 months after the last dose of investigational drug, the subject (including partner) need to have no sperm or egg donation plan or pregnancy plan and voluntarily take effective contraceptive measures.
5. Voluntarily need to sign the informed consent form before the trial, and fully understand the content, process and possible adverse reactions of the trial.

Exclusion Criteria:

1. Medical history of cardiovascular and respiratory system (such as sleep apnea syndrome, pulmonary heart disease or chronic bronchial asthma), liver, kidney, nervous system (such as epilepsy), blood system or mental disorders that the researcher considers clinically significant;
2. Medical history of cardiovascular system disease, including but not limited to history or family history of syncope, coronary heart disease (such as coronary angiography diagnosis of coronary heart disease, history of acute coronary syndrome, history of myocardial infarction, etc.), valvular heart disease, heart failure, history of non-drug-induced bradyarrhythmia, frequent ventricular premature beats, ventricular tachycardia, etc.; or previous QTc prolongation or other risk factors for torsades de pointes (hypokalemia, etc.), or a family history of a first-degree relative (i.e., biological parent, brother, sister or child) with short QT syndrome, long QT syndrome, sudden death of unknown cause in his youth (less than/equal to 40 years old), drowning or sudden infant death syndrome;
3. Medical history of symptomatic head trauma;
4. History of frequent nausea or vomiting of any etiology;
5. Medical history of glaucoma or any condition affecting pupil size;
6. Major surgery or major trauma within 6 months prior to screening or planning to undergo surgery during the study;
7. Known to be allergic to two or more kinds of food and drugs;
8. Known to be allergic to opioids, or have contraindications for the use of such drugs;
9. Difficulties in collecting venous blood, or the cases with known needle and blood sickness history;
10. Female subjects who are lactating, pregnant, preparing for pregnancy or have the abnormal pregnancy test results with clinical significance at screening;
11. Clinically significant abnormal ECG findings at screening, such as QTcF ≥ 450 ms in men and QTcF ≥ 470 ms in women; PR interval ≥ 200 ms; QRS complex duration ≥ 120 ms;
12. Abnormal vital signs at screening (systolic blood pressure < 90 mmHg or > 140 mmHg, diastolic blood pressure < 50 mmHg or > 90 mmHg; respiratory < 16 breaths/min or > 20 breaths/min; pulse < 60 beats/min or >100 beats/min) or clinically significant abnormal physical examination, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function), chest anteroposterior view or CT, abdominal color ultrasound (subject to the judgment of clinicians);
13. Subjects having clinically significant abnormalities in any of hepatitis B virus surface antigen, Treponema pallidum-specific antibody, human immunodeficiency virus antibody and hepatitis C virus antibody at screening;
14. Serum potassium, magnesium and calcium exceeding the upper limit of normal reference range or lower limit of normal reference range at screening;
15. Oxygen saturation less than 95% at screening;
16. History of any drug abuse within 1 year before screening or positive urine drug test results during screening;
17. Regular drinkers within 6 months prior to screening (drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits 40% or 150 mL of wine) or breath alcohol test results > 0 mg/100 mL, or having taken any products containing alcohol within 48 hours prior to the first use of investigational drug or not agreeing to refrain from taking any products containing alcohol during the trial;
18. Smoking more than 5 cigarettes a day within 3 months before screening, or using tobacco products within 48 hours before the first use of investigational drug, or not stopping using any tobacco products during the trial;
19. Blood donation or massive blood loss (blood loss > 400 mL, excluding female menstrual blood loss), receiving blood transfusion or using blood products within 3 months before screening;
20. Participation in any clinical trial within 3 months prior to screening;
21. Attenuated/DNA nucleic acid/recombinant protein vaccination within 4 weeks prior to screening, or inactivated vaccination within 2 weeks prior to screening, or any planned vaccination during the trial;
22. Any proposed combination of drugs that alter hepatic CYP2C9 and CYP3A4 enzyme activities, including potent inhibitors and inducers of enzymes that affect hepatic metabolism or that result in QT/QTc prolongation, 28 days prior to screening or during the trial;
23. Subjects who have used or are using opioids within 14 days before the first use of investigational drug;
24. Receiving other prescription or over-the-counter medications considered by the investigator to affect the results of this study evaluation within 14 days prior to the first dose of investigational drug;
25. Consumption of grapefruit or grapefruit juice or any food or beverage containing grapefruit within 7 days before the first dose of investigational drug, or disagreement to refrain from consumption of such food or beverage during the trial;
26. Taking or having taken any medication affecting pupil size within 48 hours prior to the first dose of investigational product;
27. Taking any caffeine-rich food or beverage (coffee, tea, cola, chocolate, etc.) within 48 hours before the first dose of investigational product, or disagreeing to refrain from consuming them during the trial;
28. Subjects who, in the opinion of the investigator, are not suitable for participation in this clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Part A： From Day 1 to Day 5 Part B： From Day 1 to Day 17
Incidence of participants with clinical laboratory abnormalities | Part A： From Day 1 to Day 5 Part B： From Day 1 to Day 17
Incidence of participants with vital signs abnormalities | Part A： From Day 1 to Day 5 Part B： From Day 1 to Day 17
Incidence of participants with physical exam abnormalities | Part A： From Day 1 to Day 5 Part B： From Day 1 to Day 17
Cmax | Pre-dose to 72h post-dose
  Cmax is defined as the observed maximum plasma concentration.
AUCinf | Pre-dose to 72h post-dose
  AUCinf is defined as the area under the plasma concentration-time curve extrapolated to infinity from time zero.
AUC0-24h | Pre-dose to 72h post-dose
  AUC0-24h is defined as the area under the plasma concentration-time curve from time zero to 24h.
AUC0-t | Pre-dose to 72h post-dose
  AUC0-24h is defined as the area under the plasma concentration-time curve from time zero to the last observable concentration.
t1/2z | Pre-dose to 72h post-dose
  t1/2z is defined as the elimination half-life.
Tmax | Pre-dose to 72h post-dose
  Tmax is defined as the observed time to reach Cmax.
CL | Pre-dose to 72h post-dose
  CL is defined as the clearance.
Vz | Pre-dose to 72h post-dose
  V is defined as the apparent volume of distribution.
MRT | Pre-dose to 72h post-dose
  MRT is defined as the mean residence time.
Ae0-t | Pre-dose to 72h post-dose
  Ae0-t is defined as the cumulative amount of drug excreted in urine or fecal from time zero to the last observable concentration.
Cumulative excretion percentage of drug through urine and feces | Pre-dose to 72h post-dose

SECONDARY OUTCOMES:
Pupil diameter | Pre-dose to 12h post-dose
Change from baseline of QTcF by timepoint | Pre-dose to 24h post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Third Hospital, Central South University, Changsha, China